CLINICAL TRIAL: NCT05208931
Title: Development of an Algorithm for Predicting Anatomical and Functional the Results of Therapy With Angiogenesis Inhibitors in Patients With Retinal Pigment Epithelium Detachments in Neovascular Age-related Macular Degeneration, Based on Primary Optical Coherence Tomography of the Macular Zone and Clinical Data.
Brief Title: Development of an Optimal Algorithm for the Management of Patients With Retinal Pigment Epithelium Detachment in Neovascular Age-related Macular Degeneration Using Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Viktoria Myasnikova, Deputy Director for Research, The S.N. Fyodorov Eye Microsurgery State Institution
Other Study IDs: 1
Record Dates: First submitted 2022-01-05; First posted 2022-01-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Machine learning; Artificial intelligence; anti-VEGF therapy; AMD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- adhesion: the group in which the adhesion of neuroepithelial detachment was observed after Anti-vascular endothelial growth factor therapy
  Interventions: Procedure: Anti-vascular endothelial growth factor therapy
- no adhesion: group in which there was no adherence of neuroepithelial detachment after Anti-vascular endothelial growth factor therapy
  Interventions: Procedure: Anti-vascular endothelial growth factor therapy
- разрыв: group in which neuroepithelial detachment rupture was observed after anti-vascular endothelial growth factor therapy
  Interventions: Procedure: Anti-vascular endothelial growth factor therapy

INTERVENTIONS:
Procedure: Anti-vascular endothelial growth factor therapy — 0.05 ml anti-VEGF, intravitreal, monthly
  Other Names: anti-VEGF

SUMMARY:
The study involves the development of an algorithm for predicting anatomical and functional results of therapy with angiogenesis inhibitors in patients with retinal pigment epithelium detachments in neovascular age-related macular degeneration, based on primary optical coherence tomography of the macular zone and clinical data.

DETAILED DESCRIPTION:
Patients were divided into 3 groups according to the results of therapy: adhesion of detachment, lack of adherence to detachment, rupture of detachment. For these groups, OCT images of the macular zone with maximum detachment before therapy are selected. These images, along with other clinical parameters, are input to the algorithm. The result is one of the 3 treatment outcomes listed above. The methods that will be used to develop the algorithm include methods for processing and transforming data, deep machine learning, metrics for calculating the accuracy of algorithms.

ELIGIBILITY:
Inclusion criteria:

* Linear B - scan through the macular area with the longest detachment
* Other pathologies

Exclusion criteria:

* Images without detachment
* Images on which it is possible to diagnose the need for therapy only in the presence of additional factors not considered in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with retinal pigment epithelium detachments with age-related neovascular macular degeneration
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Prediction algorithm | 1.09.2022
  Neural network classifier

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Myasnikova, D.Med.Sc., Study Director — Deputy Director for Research
Locations (1):
- The S.N. Fyodorov Eye Microsurgery State Institution, Krasnodar, Russia

REFERENCES:
- [Background] Rohm M, Tresp V, Muller M, Kern C, Manakov I, Weiss M, Sim DA, Priglinger S, Keane PA, Kortuem K. Predicting Visual Acuity by Using Machine Learning in Patients Treated for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2018 Jul;125(7):1028-1036. doi: 10.1016/j.ophtha.2017.12.034. Epub 2018 Feb 14. PMID 29454659
- [Background] Prahs P, Radeck V, Mayer C, Cvetkov Y, Cvetkova N, Helbig H, Marker D. OCT-based deep learning algorithm for the evaluation of treatment indication with anti-vascular endothelial growth factor medications. Graefes Arch Clin Exp Ophthalmol. 2018 Jan;256(1):91-98. doi: 10.1007/s00417-017-3839-y. Epub 2017 Nov 10. PMID 29127485
- [Background] Schmidt-Erfurth U, Bogunovic H, Sadeghipour A, Schlegl T, Langs G, Gerendas BS, Osborne A, Waldstein SM. Machine Learning to Analyze the Prognostic Value of Current Imaging Biomarkers in Neovascular Age-Related Macular Degeneration. Ophthalmol Retina. 2018 Jan;2(1):24-30. doi: 10.1016/j.oret.2017.03.015. Epub 2017 May 31. PMID 31047298
- [Background] Bogunovic H, Montuoro A, Baratsits M, Karantonis MG, Waldstein SM, Schlanitz F, Schmidt-Erfurth U. Machine Learning of the Progression of Intermediate Age-Related Macular Degeneration Based on OCT Imaging. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO141-BIO150. doi: 10.1167/iovs.17-21789. PMID 28658477
- [Background] Schmidt-Erfurth U, Waldstein SM, Klimscha S, Sadeghipour A, Hu X, Gerendas BS, Osborne A, Bogunovic H. Prediction of Individual Disease Conversion in Early AMD Using Artificial Intelligence. Invest Ophthalmol Vis Sci. 2018 Jul 2;59(8):3199-3208. doi: 10.1167/iovs.18-24106. PMID 29971444
- [Background] Kozina, E. V., S. N. Sakhnov, V. V. Myasnikova, E. V. Bykova, and L. E. Aksenova. 2021. 'Modern Trends in Diagnostics and Prediction of Results of Anti-Vascular Endothelial Growth Factor Therapy of Pigment Epithelial Detachment in Neovascular Agerelated Macular Degeneration Using Deep Machine Learning Method (Literature Review)'. Acta Biomedica Scientifica 6 (6-1): 190-203. https://doi.org/10.29413/ABS.2021-6.6-1.22.